CLINICAL TRIAL: NCT07193043
Title: A Pilot Randomized Controlled Trial of the Body Image Program (BIP) for Eating Disorder Prevention in Female University Students in Northeastern Mexico
Brief Title: Pilot Trial of the Body Image Program to Prevent Eating Disorders in Female University Students in Mexico
Acronym: Pilot-BIP-MX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Comenzar de Nuevo, AC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BIP-MX-Pilot-2025
Record Dates: First submitted 2025-09-16; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Eating Disorders; Body Dissatisfaction
Keywords: Eating Disorders Prevention; Body Image Program (BIP); Body Dissatisfaction; Dissonance-Based Intervention; Pilot Randomized Controlled Trial; University Students
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: Two-arm parallel assignment pilot randomized controlled trial, with participants allocated in a 1:1 ratio to the intervention (BIP) or waitlist control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Body Image Program (BIP) Intervention (Experimental): Participants in this arm will receive the Body Image Program (BIP), a culturally adapted, dissonance-based group intervention derived from the Body Project. The program consists of two 120-minute sessions delivered in small groups of 7-10 participants, once per week for two consecutive weeks. Sessions include verbal, written, and behavioral exercises designed to reduce thin-ideal internalization, challenge sociocultural appearance pressures, and promote positive body image. Each session concludes with homework assignments, and a commitment task is submitted within one week after Session 2.
  Interventions: Behavioral: Body Image Program (BIP)
- Waitlist Control (No Intervention): Participants in this arm will not receive the Body Image Program (BIP) during the main study period. They will complete the same assessments as the intervention group at baseline (T1), post-intervention (T2), and 4-week follow-up (T3). After the final follow-up assessment (week 6), they will be offered the opportunity to participate in the BIP between weeks 6 and 8, ensuring post-trial access in line with ethical standards.

INTERVENTIONS:
Behavioral: Body Image Program (BIP) — The Body Image Program (BIP) is a culturally adapted, dissonance-based group intervention derived from the Body Project. It is delivered in two weekly sessions of 120 minutes each, in small groups of 7-10 participants, by trained health professionals with experience in eating disorders. Activities include verbal, written, and behavioral exercises to critique sociocultural appearance ideals, reduce thin-ideal internalization, and promote more adaptive body image. Each session ends with homework: after Session 1, tasks include a behavioral challenge and reflective writing; after Session 2, a commitment activity (e.g., self-affirmation or body activism) is completed within one week and submitted by email. Participants in the waitlist control arm complete the same assessments but receive the BIP between weeks 6 and 8, after the final follow-up.
  Arms: Body Image Program (BIP) Intervention

SUMMARY:
The goal of this clinical trial is to examine whether the Body Image Program (BIP), a group workshop, is feasible and acceptable to deliver to young women in Mexico. The program is designed to help participants critically evaluate social pressures to be thin and to support healthier body attitudes.

The main questions are:

* Can the investigators successfully recruit, retain, and engage university students in the program?
* Do participants find the program useful and clear?
* Does the program show early indications of lowering body dissatisfaction and unhealthy eating attitudes?

Participants will:

* Attend 2 group sessions, one per week, each lasting approximately 2 hours (120 minutes).
* Complete short activities and homework exercises between sessions, such as reflective writing or self-affirmation tasks.
* Complete questionnaires at baseline, immediately after the program, and at 1-month follow-up.

DETAILED DESCRIPTION:
This study is a pilot randomized controlled trial designed to test the Body Image Program (BIP) with female university students in northeastern Mexico. Eating disorders and body dissatisfaction are common among young women and often begin during the university years. Most prevention programs have been evaluated only in Western countries. This study will evaluate whether the BIP, adapted for Mexico, is practical and acceptable to deliver in this setting.

The Body Image Program is a dissonance-based group intervention that encourages participants to challenge cultural pressures for thinness and to build healthier body image attitudes. In this study, participants in the intervention group will attend two sessions, each 120 minutes in duration, held once per week. Each session will include group discussions and exercises, and participants will complete short homework assignments between sessions. Sessions will be led by trained health professionals with experience in eating disorders.

A total of 30 students will be recruited and randomly assigned to either the intervention group or a waitlist control group. The intervention group will be divided into small groups of about 7-8 participants to maintain interactive discussions. Students in the waitlist control group will be offered the program after the final follow-up assessment.

The main outcomes of this study are feasibility and acceptability, including the number of eligible students who consent to participate, the proportion who complete both sessions and assessments, and whether participants find the program useful and relevant. Questionnaires will also assess body dissatisfaction, eating disorder symptoms, body appreciation, social physique anxiety, thin-ideal internalization, and appearance-based social comparisons. Assessments will take place at baseline, immediately after the program, and at 1-month follow-up.

This pilot study will provide information about whether the Body Image Program can be delivered effectively in Mexican universities and will inform the design of a larger clinical trial in the future.

ELIGIBILITY:
Inclusion Criteria:

* Female undergraduate students
* Age 18-25 years
* Currently enrolled at participating universities in northeastern Mexico
* Able to provide written informed consent
* Sufficient Spanish language proficiency to complete the intervention and assessments

Exclusion Criteria:

* Current diagnosis of a severe eating disorder requiring specialized treatment
* Current engagement in intensive psychiatric or psychological treatment
* Insufficient availability to attend the two scheduled intervention sessions

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Eating Disorder Symptoms (ED-15 Total Score) | Baseline (Week 0), Post-Intervention (Week 2), and 4-Week Follow-Up (Week 6)
  Change in eating disorder symptoms measured by the Eating Disorder-15 (ED-15; Eating Disorder-15 Questionnaire), a 15-item self-report instrument that assesses core eating disorder symptoms over the past week. Items are rated on a 0-6 Likert scale. Scores yield two subscales (Eating Concerns; Weight/Shape Over-evaluation) and a total score calculated as the mean of all items. Possible scores range from 0 to 6, with higher scores indicating greater eating disorder symptom severity.

SECONDARY OUTCOMES:
Body Dissatisfaction (BSQ-8) | Baseline (Week 0), Post-Intervention (Week 2), and 4-Week Follow-Up (Week 6)
  Body Shape Questionnaire-8 item (self-report). Total score (8-48); higher scores indicate greater body dissatisfaction.
Body Appreciation (BAS-2) | Baseline (Week 0), Post-Intervention (Week 2), and 4-Week Follow-Up (Week 6)
  ody Appreciation Scale-2 (self-report, 10 items). Scores range from 1 to 5; higher scores indicate greater body appreciation.
Social Physique Anxiety (SPAS) | Baseline (Week 0), Post-Intervention (Week 2), and 4-Week Follow-Up (Week 6)
  Social Physique Anxiety Scale-7 (self-report, 7 items). Scores range from 1 to 5; higher scores indicate greater anxiety about appearance in social settings.
Internalization of Sociocultural Ideals (SATAQ-4) | Baseline (Week 0), Post-Intervention (Week 2), and 4-Week Follow-Up (Week 6)
  Internalization of Sociocultural Ideals (Thin-Ideal Internalization Subscale of the Sociocultural Attitudes Toward Appearance Questionnaire-4) Self-report, 5 items. Each item rated on a 1-5 Likert scale. Total score is calculated as the mean of all items, with possible values ranging from 1 to 5. Higher scores indicate stronger internalization of thinness ideals.

OTHER OUTCOMES:
Recruitment Rate | During the active recruitment period, up to first participant enrollment.
  Proportion of eligible students who consent and are randomized (feasibility indicator; target ≥70%)
Retention Rate | T2 (week 2) and T3 (week 6)
  Proportion of randomized participants who complete T2 and T3 assessments (feasibility indicator; target ≥80%)
Session Adherence | Across the 2-week intervention period.
  Attendance categorized per participant as full (2/2 sessions), partial (1/2), or none (0/2); target ≥70% full adherence.
Acceptability (Participant Satisfaction) | T2 (post-intervention, week 2)
  Brief ad hoc survey developed for this study. Three single-item questions assess perceived usefulness, clarity, and relevance of the program. Each item will be summarized descriptively as mean ratings and percentage of favorable responses. No standardized scale is used.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Trujillo-ChiVacuán, MD, Principal Investigator — Comenzar de Nuevo, AC
Locations (1):
- Comenzar de Nuevo, A.C., Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including baseline characteristics and outcome measures (ED-15, BSQ-8, BAS-2, SPAS-7, SATAQ-4, PACS), will be shared. The dataset will exclude all personal identifiers and will be available together with the statistical code used for analyses.

REFERENCES:
- [Background] van Hoeken D, Hoek HW. Review of the burden of eating disorders: mortality, disability, costs, quality of life, and family burden. Curr Opin Psychiatry. 2020 Nov;33(6):521-527. doi: 10.1097/YCO.0000000000000641. PMID 32796186
- [Background] Cabassa LJ, Baumann AA. A two-way street: bridging implementation science and cultural adaptations of mental health treatments. Implement Sci. 2013 Aug 19;8:90. doi: 10.1186/1748-5908-8-90. PMID 23958445
- [Background] Shaw H, Stice E. The implementation of evidence-based eating disorder prevention programs. Eat Disord. 2016;24(1):71-8. doi: 10.1080/10640266.2015.1113832. Epub 2015 Dec 9. No abstract available. PMID 26650961
- [Background] Tavolacci MP, Grigioni S, Richard L, Meyrignac G, Dechelotte P, Ladner J. Eating Disorders and Associated Health Risks Among University Students. J Nutr Educ Behav. 2015 Sep-Oct;47(5):412-20.e1. doi: 10.1016/j.jneb.2015.06.009. PMID 26363936
- [Background] Villalobos-Hernandez A, Bojorquez-Chapela I, Hernandez-Serrato MI, Unikel-Santoncini C. Prevalencia de conductas alimentarias de riesgo en adolescentes mexicanos: Ensanut Continua 2022. Salud Publica Mex. 2023 Jun 12;65:s96-s101. doi: 10.21149/14800. Spanish. PMID 38060957
- [Background] Trujillo-ChiVacuan E, Winterman-Hemilson B, Compte EJ, Rodriguez G, Perez M, Black Becker C. Adaptation and implementation of body project as a universal body image program in Mexico and Latin America. Eat Disord. 2024 Nov-Dec;32(6):644-665. doi: 10.1080/10640266.2024.2360256. Epub 2024 Jun 3. PMID 38828520
- [Background] Fairburn CG, Cooper Z, Shafran R. Cognitive behaviour therapy for eating disorders: a "transdiagnostic" theory and treatment. Behav Res Ther. 2003 May;41(5):509-28. doi: 10.1016/s0005-7967(02)00088-8. PMID 12711261
- [Background] Stice E, Yokum S, Waters A. Dissonance-Based Eating Disorder Prevention Program Reduces Reward Region Response to Thin Models; How Actions Shape Valuation. PLoS One. 2015 Dec 7;10(12):e0144530. doi: 10.1371/journal.pone.0144530. eCollection 2015. PMID 26641854
- [Background] Stice E, Rohde P, Gau J, Shaw H. An effectiveness trial of a dissonance-based eating disorder prevention program for high-risk adolescent girls. J Consult Clin Psychol. 2009 Oct;77(5):825-34. doi: 10.1037/a0016132. PMID 19803563
- [Derived] Trujillo-ChiVacuan EM, Winterman-Hemilson B, Trujillo-Valdes EY, Cortes-Morales A, Compte EJ. Culturally adapted body image program for Mexican university women: feasibility, acceptability, and cultural relevance in a Pilot RCT protocol. Front Psychiatry. 2026 Jan 14;16:1717786. doi: 10.3389/fpsyt.2025.1717786. eCollection 2025. PMID 41614095